CLINICAL TRIAL: NCT01755351
Title: Comparative Study About the Influence of Diabetes Diatress and Depression on Treatment Adherence in Chinese Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, cuiping-xu, Qianfoshan Hospital, Shandong Provincial Hospital
Other Study IDs: ShandongPH
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Compare Diabetes Distress and Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
An effective treatment adherence was a key to make the treatment success, some reports had shown that psychologicl factors impact patients adherence seriously,however, in China, the researches were only limited to depression and diabetes,diabetes distress was neglected. Some western studies had demonstrated the impact of diabetes distress on diabetes. Thus, we hypothesized that: 1.perhaps our present depression-oriented health education was inadequate to promote patients' adherence, diabetes distress might played a more important part than depression in patients' treatment adherence. 2. there might be a high prevalence of diabetes distress in Chinese type 2 diabetes; so, the comparative study between diabetes distress and depresion was conducted.

Objectives: to explore the relationship of diabetes-related distress and depression，and to compare the influence of diabetes distress and depression on treatment adherence in Chinese type 2 diabetes .

Research design and method:we surveyed 200 type 2 diabetic patients from 2 third-class hospitals using the Diabetes Distress Scale, Zung Self-rating Depression Scale, and Revised Treatment Adherence in Diabetes Questionnaire (RADQ)simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* 1)aged between 18-80 years, 2)diagnosed with diabetes for at least 6 month, 3) having the ability to communicate fluently and clearly,

Exclusion Criteria:

* patients who had the diagnosis of dementia or psychosis and severe diabetes complications (e.g., on dialysis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetes who visited the two local hospitals between December 2011 and April 2012, were invited to participate in this cross-sectional survey study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The influence of diabetes distress on treatment sdherence | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital Shandong province, Jinan, China